CLINICAL TRIAL: NCT03294265
Title: A Peer Support Program to Enhance Treatment Adherence in Patients With Type 2 Diabetes Mellitus
Brief Title: A Peer Support Program to Enhance Treatment Adherence in Patients With Type 2 DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Carlos Aguilar, Coordinator of the Research Unit in Metabolic Diseases at the Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1853
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Peer support; WhatsApp
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Non-probabilistic sampling, by convenience (for the leaders). Randomization was performed by random stratified sampling, for which we considered age, sex and metabolic parameters (HbA1c, tryglycerides, blood pressure and body-mass index) of every patient in its fourth visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer support group (Experimental): Patients who accept to participate in the protocol and are randomized to the intervention group will be invited to five sessions, one per bimester, that will be carried out in our facilities until their next appointment to the centre (fifth visit). All of them will be coordinated by a group leader.
  Interventions are made each bimester in 2 hours in peer support sessions in which the patients discuss and reinforce the following topics: grief stages, control goals, self-care activities, adequate diet planning and diminish sedentary lifestyle.
  Interventions: Behavioral: Peer support sessions; Behavioral: Reminders
- Control group (Active Comparator): Patients who accept to participate in the protocol and are randomized to the control group will receive weekly messages and reminders about self-care to their cell phones via WhatsApp.
  Interventions are made by sending each week a self-care reminder via WhatsApp and questionnaires about self-care activities and drugs
  Interventions: Behavioral: Reminders

INTERVENTIONS:
Behavioral: Peer support sessions — Stages of mourning and motivation Patients introduce themselves, share their experience and mention a strategy on moving on to the next stage Reminder of metabolic control goals Leaders write on the board metabolic variables and ask everybody the goal values. Patients share their results and mention plans to improve them Self-care activities Leaders ask who owns a glucometer, how regularly they use it, its importance and consequences of not doing so.
  Simplified meal plan Everyone brings a snack. Leaders ask if each snack is appropriate, how everyone carries out their meal plan, barriers and possible strategies Activities to increase physical activity Everyone compares who achieves 10 thousand steps/day and who doesn't, then mention benefits of exercise
  Arms: Peer support group
Behavioral: Reminders — Creation of a group on WhatsApp to send leaders and patients a weekly reminder on the different areas of self-care, such as foot care, self-monitoring, adherence to meal plan, medication and exercise.
  This intervention will be applied to both groups.

SUMMARY:
Diabetes Mellitus (DM) affects patients' quality of life in different dimensions. Therefore, it is considered a priority to design and create specialized intervention programs in order to prevent and decrease complications. The peer support program studies have shown to Increase adherence to treatment and the proportion of patients with adequate long-term metabolic control.

The benefits that these programs bring are the social and emotional support in the daily management of the disease through shared experiences and communication in a continuous way.

There are only a few peer support programs in Mexico, thus it is required to investigate the effects of their implementation in our environment to promote empowerment and maintain long-term lifestyle changes. The present study has the objective to enhance self-care behaviors and health empowerment in patients with diabetes through peer support.

DETAILED DESCRIPTION:
The traditional model of attention has not been able to face the diabetes epidemic mainly because it is treated like an acute disease instead of like a chronic condition. Given that it requires a continuous and integrated management that cares for all the aspects of the patient's disease, it is fundamental that the patients learn to live with diabetes, and to manage it effectively to improve their life quality and reduce the risks of long term complications.

The peer support programs include people who live with the same condition (patients, relatives and friends) who have received training related to their treatment, becoming an important social, emotional and practical support in the daily care of chronic diseases.They become comfortable enough as to share their emotions and experiences with other patients with their same condition.

Many studies have shown that the patients with diabetes who commit to provide peer support to others also improve their self-care and glycemic long-term control.

The meetings with group leaders consist discussions among the patients where they share experiences and solutions to barriers.

The Center of Comprehensive Care for the Patient with Diabetes (CAIPaDi) was created with the objective of investigating about new strategies to promote empowerment, self-efficacy and the reach of metabolic control in order to prevent diabetes complications (protocol "Validation of an integrated attention model for the patient with type 2 diabetes" reference number 1198). The inclusion criteria are: less than 5 years of diagnosis of diabetes, absence of chronic complications, not smoking and having a relative to join them in all the sessions. The program consists of 4 initial visits, one per month, and includes attention from 9 specialties: endocrinology, psychology, nutrition, ophthalmology, diabetes education, odontology, physical activity, foot care and psychiatry. Upon conclusion of the fourth visit, a counter-reference of each patient is sent to their corresponding particular physician. In this report, each specialty explains in a detailed manner the strengths and opportunity areas of the patient. Afterwards, the patient is given an appointment a year after concluding the first phase of the program (visit 5) and a year after this visit (visit 6).

Description of the interventions

1. Identification of the "group leaders"

Patients who fulfill the eligibility criteria will be invited and asked to sign the informed consent, afterwards they will attend 7 training sessions of 60 minutes each, the following topics will be assessed in each of them:

1. Reinforcement of the metabolic control goals and most common problems in diabetes.
2. Self-care activities: detection and appropriate treatment of hypoglycemia, glucose self-monitoring, foot care and actions on concomitant diseases.
3. Adherence to meal plan
4. Structuration of activities to increase physical activity or diminish sedentarism and measurement methods (steps per day, identification of exercise intensity levels)
5. Emotional aspects of diabetes (duel and motivation stages)
6. Adhesion to pharmacologic treatment (medications and insulin)

Each session will be arranged by a team researcher and will be structured in the following way:

10 minutes: reminder of activities and resolution of doubts from the previous session 50 minutes: new subject of each session

After the patient has completed the training, an objective structured clinical evaluation will be performed. The patients who approve the evaluation will receive a group management session where they will obtain the necessary skills to motivate and transmit information to the rest of the group.

Phase 2: Integration of patient groups All the patients who finish the fourth visit in the centre will be invited, those who accept will be randomized into participants or control patients.

Each group will be formed by 2 group leaders and 5 patients. The minimum number of participants per session will be 2 (one leader and one patient). Five sessions are projected, one every 2 months, where the next topics will be reviewed in each of them:

1. Identification of motivation and duel stages
2. Reinforcement of metabolic control goals
3. Self-care activities:detection and appropriate treatment of hypoglycemia, glucose self-monitoring, foot care and actions on concomitant diseases and insulin application.
4. Enhancement of adhesion to simplified meal plan and recognition of portions
5. Structuration of activities to boost physical activity and/or reduce sedentarism and how to measure it (steps per day and identification of exercise intensity levels)

Motivational messages and reminders will be created and sent by WhatsApp (cross-platform instant messaging application) weekly to patients, controls and group leaders to strengthen adhesion to integral treatment.

Every session will be carried out in the facilities of the centre, where the leaders will share their experiences with the rest of the group to reinforce self-care activities.

ELIGIBILITY:
Inclusion Criteria:

* Leaders:
* Completion of the fifth visit and fulfillment of the following criteria:
* HbA1c <7%
* Triglycerides <150 mg/dl
* Non-HDL cholesterol <130 mg/dl
* Blood pressure <130/80 mmHg
* Normal weight or a reduction of 10% since the first visit
* Approval after a psychiatric and psychologic evaluation
* Patients:
* Completion of the fourth visit in the centre
* Absence of diabetes complications
* Non-smokers

Exclusion Criteria:

* Non-attendance to more than one session

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | 1 year
  A value of less than 7%

SECONDARY OUTCOMES:
Triglycerides | 1 year
  A value of less than 150 mg/dl
Blood pressure | 1 year
  A value of less than 130/80 mmHg
Non-HDL cholesterol | 1 year
  A value of less than 130 mg/dl
Weight | 15 months
  Maintenance of an appropriate weight or a 10% weight reduction in overweight or obese patients from the first to the fifth visit
Hypoglycemia events | 1 year
  Reduction of the number of hypoglycemia events
Emergency attendance | 1 year
  Reduction of the number of attendances to the emergency rooms
Foot care | 1 year
  Increase in the number of days the patients check their feet

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cristina García Ulloa, Dr., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daaleman TP, Fisher EB. Enriching Patient-Centered Medical Homes Through Peer Support. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S73-8. doi: 10.1370/afm.1761. PMID 26304975
- [Result] Ayala GX, Ibarra L, Cherrington AL, Parada H, Horton L, Ji M, Elder JP. Puentes hacia una mejor vida (Bridges to a Better Life): Outcome of a Diabetes Control Peer Support Intervention. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S9-17. doi: 10.1370/afm.1807. PMID 26304977
- [Result] de Vries L, van der Heijden AA, van 't Riet E, Baan CA, Kostense PJ, Rijken M, Rutten GE, Nijpels G. Peer support to decrease diabetes-related distress in patients with type 2 diabetes mellitus: design of a randomised controlled trial. BMC Endocr Disord. 2014 Mar 4;14:21. doi: 10.1186/1472-6823-14-21. PMID 24593296
- [Result] van Puffelen AL, Rijken M, Heijmans MJ, Nijpels G, Rutten GE, Schellevis FG. Living with diabetes: a group-based self-management support programme for T2DM patients in the early phases of illness and their partners, study protocol of a randomised controlled trial. BMC Health Serv Res. 2014 Apr 1;14:144. doi: 10.1186/1472-6963-14-144. PMID 24690511
- [Result] Fisher EB, Ayala GX, Ibarra L, Cherrington AL, Elder JP, Tang TS, Heisler M, Safford MM, Simmons D; Peers for Progress Investigator Group. Contributions of Peer Support to Health, Health Care, and Prevention: Papers from Peers for Progress. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S2-8. doi: 10.1370/afm.1852. PMID 26304968
- [Result] Ghorob A, Vivas MM, De Vore D, Ngo V, Bodenheimer T, Chen E, Thom DH. The effectiveness of peer health coaching in improving glycemic control among low-income patients with diabetes: protocol for a randomized controlled trial. BMC Public Health. 2011 Apr 1;11:208. doi: 10.1186/1471-2458-11-208. PMID 21457567
- [Result] Goldman ML, Ghorob A, Eyre SL, Bodenheimer T. How do peer coaches improve diabetes care for low-income patients?: a qualitative analysis. Diabetes Educ. 2013 Nov-Dec;39(6):800-10. doi: 10.1177/0145721713505779. Epub 2013 Oct 29. PMID 24168838
- [Result] Knox L, Huff J, Graham D, Henry M, Bracho A, Henderson C, Emsermann C. What Peer Mentoring Adds to Already Good Patient Care: Implementing the Carpeta Roja Peer Mentoring Program in a Well-Resourced Health Care System. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S59-65. doi: 10.1370/afm.1804. PMID 26304973
- [Result] Murray NJ, Gasper AV, Irvine L, Scarpello TJ, Sampson MJ. A motivational peer support program for type 2 diabetes prevention delivered by people with type 2 diabetes: the UEA-IFG feasibility study. Diabetes Educ. 2012 May-Jun;38(3):366-76. doi: 10.1177/0145721712440332. Epub 2012 Apr 6. PMID 22491396